CLINICAL TRIAL: NCT06546176
Title: Comparative Study Between End to End Anastomosis With Omega Suture Versus End to Anterior Rectal Wall In Colorectal Anastomosis in Sigmoid and Upper Rectal Cancer
Brief Title: End to End Anastomosis With Omega Suture Versus End to Anterior Rectal Wall In Colorectal Anastomosis in Sigmoid and Upper Rectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Asmaa fathi, Assistant Lecturer of General Surgery, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13/8/2023
Record Dates: First submitted 2024-08-04; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: End to End Anastomosis; Colorectal Anastomosis; End to Anterior Rectal Wall; Sigmoid Cancer; Upper Rectal Cancer
MeSH Terms: conditions — Sigmoid Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A(end to end with Omega suture) (Other): After the rectum was divided with a linear stapler, the circular stapler was placed allowing the anvil rod to penetrate the rectal stump near the linear stapler line. An omega suture including both ends of the linear stapler line was placed. The linear stapler line was approximated around the anvil rod of the circular stapler in an omega shape fashion as the omega suture was tied. This technique resulted in a complete resection of linear stapler line by the circular stapler.
  Interventions: Other: End to end with Omega suture
- Group B (end to anterior rectal wall) (Other): A burse string suture was applied over the anvil of the circular stapler at the transection point of the descending colon using prolene 2/0.
  The circular stapler introduced though the anus and its rod directed toward the anterior rectal wall and colorectal anastomosis was performed.
  Interventions: Other: End to anterior rectal wall

INTERVENTIONS:
Other: End to end with Omega suture — After the rectum was divided with a linear stapler, the circular stapler was placed allowing the anvil rod to penetrate the rectal stump near the linear stapler line. An omega suture including both ends of the linear stapler line was placed. The linear stapler line was approximated around the anvil rod of the circular stapler in an omega shape fashion as the omega suture was tied. This technique resulted in a complete resection of linear stapler line by the circular stapler.
  Arms: Group A(end to end with Omega suture)
Other: End to anterior rectal wall — A burse string suture was applied over the anvil of the circular stapler at the transection point of the descending colon using prolene 2/0.
  The circular stapler introduced though the anus and its rod directed toward the anterior rectal wall and colorectal anastomosis was performed.
  Arms: Group B (end to anterior rectal wall)

SUMMARY:
The aim of this study is to compare end to end anastomosis with omega suture versus end to anterior rectal wall in colorectal anastomosis as regard post operative anastomotic leakage, bowel function, operative time and intra operative blood loss.

DETAILED DESCRIPTION:
Colorectal cancer has been reported to be the 3rd most common and the second most deadly cancer world wide.

Anterior resection is the gold standard operation for both rectal and recto-sigmoid cancer with considering oncological safety maintenance to be the most important goal which can be achieved by keeping abundant resection margin and ensuring anastomotic safety, despite the technical difficulties of working in a narrow deep pelvis.

Understanding the characteristics of each anastomotic technique and establishing a stable anastomotic procedure both are pillars in anastomotic leakage prevention.

The intersection of the linear staple line and circular staple line in conventional anastomotic way is considered a risk factor for anastomotic leakage by creating stapled corners (called "dog-ears") which considered potentially ischemic and represent the area with high incidence of anastomotic leakage. Single stapled technique using ether end to end with omega suture or end to side stapled anastomosis allows avoidance of the formation of this intersection.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years.
* Both sexes.
* Recto sigmoidal carcinoma.
* Upper rectal cancer.

Exclusion Criteria:

* Patients younger than 18 years
* Recurrent or non-resectable cancer
* Complicated cancer (e.g., obstructed or perforated)
* Previous left-sided colorectal surgery or anorectal surgeries
* Lower rectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage | 5 days after surgery
  Anastomotic leakage will be measured for 5 days after surgery

SECONDARY OUTCOMES:
Operative time | Until the procedure is completed
  Operative time will be measured from the start of surgery till the end of surgery.
Hospital stay | 28 days postoperative
  Hospital stay will be assessed from admission till discharge from hospital
Time of bowel function | 7 days postoperative
  Time of bowel function will be assessed
Wound complications | 7 days postoperative
  Wound complications will be recorded as bleeding and infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.